**Independent Ethics Committee** 

**IRCCS Humanitas Clinical Institute** 

Rozzano, 29/06/2023

Subject: "Preimplantation genetic testing for monogenic disease: the experience of a single center."

This Ethics Committee is hereby notified of the retrospective work with the above title.

The Principal Investigator Prof.Paolo Emanuele Levi-Setti declares that the treatment under study is part of Good Clinical Practice and that nothing is performed unless required by the normal clinical diagnostic course of the patients.

Sincerely,

Paolo Emanuele Levi-Setti, MD

Humanitas Research Hospital

Director and Chair, Department of Gynecology, Division of Gynecology and Reproductive Medicine, Humanitas Fertility Center

do to Cen Sles

EBCOG/ ESHRE European Center in Reproductive Medicine

Professor (Adjunct) of Obstetrics, Gynecology and Reproductive Science. Yale University, School of Medicine.